CLINICAL TRIAL: NCT00390520
Title: A Single-center, Double-blind, Randomized, Placebo-controlled, Cross-over Study to Assess the Effect of Vildagliptin on Glucagon Counterregulatory Response During Hypoglycemia in Patients With Type 2 Diabetes.
Brief Title: Efficacy and Safety of Vildagliptin Versus Placebo in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2386
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2009-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin; glucagon; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
This mechanistic study is designed to investigate the effect of vildagliptin on the sensitivity of the a-cell to glucose under hypoglycemic conditions in patients with type 2 diabetes (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM, diagnosed at least 6 weeks prior to visit 1, who have had no treatment with oral antidiabetic agents for at least 12 weeks prior to study entry (visit 1) and no treatment with oral antidiabetic agents at any time in the past for > 3 consecutive months
* >/= 18 years
* Body mass index in the range of 22-35 kg/m2
* HbA1c </=7.5%

Exclusion Criteria:

* Type 1 diabetes
* Acute metabolic diabetic complications
* Evidence of significant diabetic complications
* Insulin treatment within the past 6 months

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Glucagon counterregulatory response to hypoglycemia of the last 30 min of the 2.5 mM hypoglycemic clamp after 4 weeks treatment

SECONDARY OUTCOMES:
Glucagon counterregulatory response to hypoglycemia assessed as glucagon Cmax of the 2.5 mM hypoglycemic clamp step after 4 weeks treatment
The 'insulin secretion rate relative to glucose' at the hypoglycemic clamp step after 4 weeks treatment
Change from baseline on hemoglobinA1c (HbA1c)and fasting plasma glucose
Safety based primarily on frequency of adverse events, number of notable abnormal laboratory values, and frequency and severity of hypoglycemic events

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Basel, Switzerland

REFERENCES:
- [Derived] Ahren B, Schweizer A, Dejager S, Dunning BE, Nilsson PM, Persson M, Foley JE. Vildagliptin enhances islet responsiveness to both hyper- and hypoglycemia in patients with type 2 diabetes. J Clin Endocrinol Metab. 2009 Apr;94(4):1236-43. doi: 10.1210/jc.2008-2152. Epub 2009 Jan 27. PMID 19174497